CLINICAL TRIAL: NCT06090656
Title: Bevacizumab in Combination With Sintilimab Versus Transcatheter Arterial Chemoembolization for the Treatment of Intermediate Stage Hepatocellular Carcinoma (Beyond Up-To-Seven Criteria), A Prospective, Randomized, Controlled Clinical Trial
Brief Title: Bevacizumab in Combination With Sintilimab Versus Transcatheter Arterial Chemoembolization for the Treatment of Intermediate Stage Hepatocellular Carcinoma (Beyond Up-To-Seven Criteria)
Acronym: BEST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Binkui Li, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2022-759-01
Record Dates: First submitted 2023-10-14; First posted 2023-10-19 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab combined with Sintilimab (Active Comparator): Bevacizumab combined with sintilimab, sindilizumab 200 mg IV d1, Q3W, combined with bevacizumab 15 mg/kg IV d1, Q3W treatment, treatment continued until disease progression, development of intolerable toxic reactions
  Interventions: Drug: Bevacizumab combined with Sintilimab
- Transcatheter arterial chemoembolization (Sham Comparator): Transcatheter arterial chemoembolization, patients were treated with cTACE, and the efficacy was assessed by repeat CT/MRI 1 month after the initial treatment, and if the tumor still had arterial phase enhancement, TACE treatment could be supplemented until treatment failure and withdrawal of consent.
  Interventions: Procedure: Transcatheter arterial chemoembolization

INTERVENTIONS:
Drug: Bevacizumab combined with Sintilimab — Bevacizumab combined with sintilimab, sindilizumab 200 mg IV d1, Q3W, combined with bevacizumab 15 mg/kg IV d1, Q3W treatment, treatment continued until disease progression, development of intolerable toxic reactions
  Arms: Bevacizumab combined with Sintilimab
Procedure: Transcatheter arterial chemoembolization — Transcatheter arterial chemoembolization, patients were treated with cTACE, and the efficacy was assessed by repeat CT/MRI 1 month after the initial treatment, and if the tumor still had arterial phase enhancement, TACE treatment could be supplemented until treatment failure and withdrawal of consent.
  Arms: Transcatheter arterial chemoembolization

SUMMARY:
Transcatheter arterial chemoembolization (TACE) is recommended as the standard of care for patients with intermediate-stage hepatocellular carcinoma (HCC) (i.e., BCLC stage B). However, these patients is heterogeneous in terms of liver functional, tumor size and tumor number, and not all patients with mid-stage HCC will benefit from TACE. The ORIENT-32 trial confirmed the efficacy of sintilimab in combination with bevacizumab for unresectable hepatocellular carcinoma. No study has yet explored whether this regimen is appropriate for patients with BCLC stage B. The purpose of this study is to explore whether bevacizumab in combination with sintilimab is superior to conventional TACE therapy in patients with HCC with beyond-Up-to-seven criteria.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed hepatocellular carcinoma, or meet the American Association for the Study of Liver Diseases (AASLD) clinical diagnostic criteria for hepatocellular carcinoma.

Age ≥ 18 years old. ECOG score 0. No systemic systemic antitumor therapy against hepatocellular carcinoma and transhepatic arterial intervention prior to treatment.

Tumour extent: Barcelona Clinic Liver Cancer (BCLC) stage B unsuitable for radical surgery and/or local treatment, together with a tumour load exceeding the Up-To-Seven criteria, i.e. the sum of the size (in centimetres) of the largest tumour in the liver and the number of tumours greater than 7; tumor was bilobed with multiple lesions; at least one measurable lesion with CT/MRI showing arterial phase enhancement; no portal vein thrombus; and no extrahepatic metastasis.

No risk of variceal bleeding: CT/MRI/esophagogastroduodenoscopy within 6 months did not suggest esophagogastric fundic varices and active ulcers.

Child-Push A Normal hematologic function (platelets >75×10E9/L; leukocytes >3.0×10E9/L; neutrophils >1.5×10E9/L) Serum bilirubin ≤ 1.5 times the upper limit of normal (ULN), transaminases ≤ 3 times the ULN No ascites, normal coagulation function, albumin ≥ 30g/L Serum creatinine less than 1.5 times the upper limit of normal (ULN) Life expectancy > 3 months

Exclusion Criteria:

Previously confirmed fibrous lamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, and bile duct carcinoma.

history of hepatic encephalopathy or a history of liver transplantation. pleural fluid, ascites, and pericardial effusion with clinical symptoms requiring drainage.

Acute or chronic active hepatitis B or C infection with hepatitis B virus (HBV) DNA > 2000 IU/ml or 10E4 copies/ml; hepatitis C virus (HCV) RNA > 10E3 copies/ml; positive for both hepatitis B surface antigen (HbsAg) and anti-HCV antibodies. Those who were below the above criteria after antiviral therapy could be enrolled.

had any of the following within the 12 months prior to study entry: myocardial infarction, severe/unstable angina, coronary artery bypass graft, congestive heart failure, cerebrovascular accident (including transient ischemic attack), pulmonary embolism; ongoing: arrhythmia ≥ grade 2 according to NCI-CTCAE criteria, prolonged QTc interval (>450 ms in men , women >470 ms); Uncontrollable hypertension, systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg after optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy.

Renal failure requiring hemodialysis or peritoneal dialysis; Severe dysfunction of other vital organs; History of malignancy other than hepatocellular carcinoma within 3 years prior to screening, except for malignancies with negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as adequately treated cervical carcinoma in situ, non-melanoma skin cancer, limited prostate cancer, ductal carcinoma in situ, or stage I uterine cancer; evidence of brain or soft meningeal lesions; hemophilia or bleeding tendencies, who are taking therapeutic doses of anticoagulant therapy such as coumarin derivative drugs; pregnant or lactating females, all female patients of childbearing potential must have a pregnancy test (serum or urine) within 7 days prior to enrollment and have a negative result; Prior organ transplant history; Known HIV infection; Active Tuberculosis chemotherapy drug allergy; comorbid systemic or other serious co-morbidities that, in the judgment of the investigator, would make the patient unsuitable for participation in this study or substantially interfere with the appropriate assessment of the safety and toxicity of the prescribed protocol.

Active or history of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, dry syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

Patients with other serious acute, chronic physical or psychiatric illnesses or abnormal laboratory tests that may increase the risk associated with study participation or that may interfere with the interpretation of study results or that the investigator deems unsuitable for enrollment.

Patients with any history of significant noncompliance with medical regimens or inability to obtain reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
progression free survival，PFS | 24 months
  Assessed using the mRECIST criteria, defined as patient survival without tumor progression from the start of randomization to the end of year 2

SECONDARY OUTCOMES:
overall survival, OS | 24 months
  Defined as the time from the start of randomization to death from any cause.
post-progression survival，PPS | 24 months
  Defined as overall survival minus progression-free survival time
Time to failure of treatment strategy | 24 months
  Time from randomization to death or need for further treatment options
Duration of Response, DOR | 24 months
  Time from initial response to disease progression or death in patients identified as CR or PR according to mRECIST and RECIST 1.1 criteria
objective response rate，ORR | 24 months
  Evaluated according to the criteria for evaluating efficacy in solid tumors (mRECIST and RECIST 1.1)
conversion rate to resection | 24 months
  Rate of patients whose tumors regressed and underwent surgical resection
Patient-reported outcomes, PRO | 24 months
  Change from baseline in overall health, quality of life, physical, role, emotional, and social functioning using the IL42-EORTCQLQ-C30 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China